CLINICAL TRIAL: NCT02231554
Title: Effectiveness of Feldenkrais Method Versus a Back School Program in Patients With Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Feldenkrais vs Back School for Treating Chronic Low Back Pain: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, medical director, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3297/2014
Record Dates: First submitted 2014-08-08; First posted 2014-09-04 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; quality of life; rehabilitation; exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Feldenkrais (Experimental): The Feldenkrais method is a self education method that uses the somatic sensory-motor learning to enhance the functions of people in daily life activities through the awareness of their motor habits and the experience of more efficient alternatives.
  Interventions: Other: Feldenkrais Method
- Back School (Active Comparator): The Back School teaches the patient, with theoretical and practical knowledge, how to defend his own back from the pain and how to prevent their disease, considering awareness and education as important parts of the therapeutic process .
  Interventions: Other: Back School

INTERVENTIONS:
Other: Feldenkrais Method — The program of Awareness Through Movement ® chosen for this study, teaches the basic movements of the column. The aim is to stimulate changes in the chronic pathological patterns and in the distorted kinesthetic perceptions that so often hinder the rehabilitation of chronic non-specific low back pain. The patients will be treated in outpatient with the Feldenkrais method. Each group will consist of four or five patients who carry out the rehabilitation treatment with a frequency of twice a week for five consecutive weeks for a total of 10 sessions, each lasting about one hour.
  Other Names: Awarness through movement program
  Arms: Feldenkrais
Other: Back School — The rehabilitation program of Back School is divided into two parts: one theoretical and one practical. To obtain an effective action not only in reducing pain but also in preventing relapse, the Back School acts on the typical risk factors of chronic non-specific low back pain, such as incorrect postures and movements, psychological stress, poor physical fitness, overweight, obesity, smoking, and insufficient knowledge of the spine. The patients will be treated in outpatient with a Back School program. Each group will consist of four or five patients who carry out the rehabilitation treatment with a frequency of twice a week for five consecutive weeks for a total of 10 sessions, each lasting about one hour.
  Arms: Back School

SUMMARY:
The purpose of this study study is to determine whether the Feldenkrais method is effective on pain control, functional recovery and quality of life in patients with chronic low back pain by comparing it with a Back School program.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic nonspecific low back pain for at least three months;
* Subjects aged between 18 and 80 years.

Exclusion Criteria:

* Presence of acute low back pain;
* Low back pain due to other causes (vertebral fractures, spondylolisthesis, herniated discs, lumbar canal stenosis);
* CNS and/or PNS disorders;
* Systemic inflammatory disease (eg rheumatoid arthritis);
* Systemic infectious disease;
* Neoplastic disease;
* Previous Surgery;
* Cognitive impairment;
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change of Visual analogue scale (VAS) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It is based on a ten point scale, where 0 means no pain and 10 the greatest pain ever. It enables the patients to express their pain intensity as numerical values.

SECONDARY OUTCOMES:
Change of SF-36 Health Survey Questionnaire from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  The questionnaire is divided into eight sub-categories that measure the physical activity, role limitations due to physical health and emotional state, physical pain, the perception of general health, vitality, social activities, mental health and changes in health status and two indices that summarize the overall assessment of the subject with respect to his physical health (ISF) and mental (ISM).
Change of McGill Pain Questionnaire from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  This scales evaluates the degree of functional impairment in activities of daily life caused by pain. It consist of ten sections including pain intensity, personal care, lifting, walking, sitting standing, sleeping, sex, social life and travelling. Each section includes six sentences relating to different level of limitation in the same activity (0: no limitation, 5: maximal limitation).
Change of Waddell Disability Index from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It includes nine parameters: pain experienced in a sitting position, travelling, standing,walking and lifting weights and the need to put on or remove footwear, sleep disturbance, life restriction and sex life restriction to measure. The maximum score is 9 points. A score > 5 indicates significant disability.
Change of Multidimensional Assessment of Interoceptive Awarness (MAIA) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  The questionnaire is divided into 32 items organized into eight subcategories consisting of three to seven items each. The subcategories measure: the awareness of unpleasant, pleasant or neutral body sensations, the tendency not to ignore the feelings of pain or discomfort, not to worry about painful sensations or discomfort, the ability not to draw attention away from body sensations, awareness of the existence of connections between body sensations and emotional status, the ability to control the psychological stress by focusing on body sensations, the ability to listen to your body and the belief that the experiences coming from your body are safe and reliable. It 'a multidimensional assessment questionnaire and self-administered. For each subcategory, the patient may express a score from 0 (never) to 5 (always), the highest score corresponds to a higher level of awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Maria Saraceni, Study Director — Umberto I Hospital, Sapienza University of Rome
Locations (1):
- Umberto I Hospital, Rome, Italy